CLINICAL TRIAL: NCT04601324
Title: Randomized Controlled Trial Evaluating Combination Rupatadine and Fluticasone Propionate Compared to Azelastine Hydrochloride and Fluticasone Propionate in Treating Allergic Rhinitis
Brief Title: Allergic Rhinitis Combination Pharmacotherapy Efficacy Study
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: PI did not pursue this study
Sponsor: St. Paul's Sinus Centre (Other)
Responsible Party: Principal Investigator, Dr. Andrew Thamboo, MD, Principal Investigator, St. Paul's Sinus Centre
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Allergic Rhinitis Protocol
Record Dates: First submitted 2020-10-19; First posted 2020-10-23 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2023-10

CONDITIONS: Allergic Rhinitis
Keywords: Allergic Rhinitis; Oral Antihistamine; Nasal Steroid; Nasal Antihistamine Spray
MeSH Terms: conditions — Rhinitis, Allergic | interventions — Fluticasone; azelastine; rupatadine

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Dymista (Azelastine hydrochloride and fluticasone propionate) (Active Comparator): Participants will receive standard of care, which includes twice daily MP-AzeFlu nasal spray (formulation of 137 mg of azelastine hydrochloride and 50 mcg of fluticasone propionate per spray) separated by 12 hours.
  Interventions: Drug: Azelastine hydrochloride and fluticasone propionate
- Fluticasone Propionate and Rupatadine (Experimental): Participants will administer fluticasone propionate nasal spray once daily (2 sprays in each nostril, 50 mcg fluticasone propionate per spray)and 1 tablet of Rupatadine (10mg) once daily in the morning.
  Interventions: Drug: Fluticasone Propionate; Drug: Rupatadine

INTERVENTIONS:
Drug: Fluticasone Propionate — Participants will be required to use fluticasone propionate nasal spray twice daily.
  Other Names: Flonase
  Arms: Fluticasone Propionate and Rupatadine
Drug: Azelastine hydrochloride and fluticasone propionate — Participants will be required to administer twice daily MP-AzeFlu nasal spray (formulation of 137 mg of azelastine hydrochloride/50 mg of fluticasone propionate) separated by 12 hours.
  Other Names: Dymista
  Arms: Dymista (Azelastine hydrochloride and fluticasone propionate)
Drug: Rupatadine — Rupatadine once daily for a total of 2 weeks.
  Other Names: RUPALL
  Arms: Fluticasone Propionate and Rupatadine

SUMMARY:
Combination pharmacotherapy is often used in people who have failed mono-therapies in managing their bothersome allergic rhinitis symptoms . However, there is a paucity of research indicating the most effective combination therapies in managing allergic rhinitis. This study aims to evaluate the efficacy of oral antihistamine (rupatadine) combined with nasal steroid (fluticasone propionate) compared to a well-studied combination therapy of nasal steroid with nasal antihistamine spray (MP-AzeFlu).

DETAILED DESCRIPTION:
Allergic rhinitis is a common inflammatory disorder of the nose that is increasing in prevalence worldwide. Symptoms of allergic rhinitis has a significant negative impact on an individual's quality of life. When the symptoms are not well managed with allergen avoidance and first line pharmacotherapies, patients often resort to using a combination of medications. Physicians may recommend combination therapies to patients with moderate-to-severe allergic rhinitis, however, there is a scarcity of research indicating efficacy of combination therapy use. The investigators of this study aim to evaluate the efficacy of combining oral antihistamine (rupatadine) with nasal steroid (fluticasone propionate) compared to a well-studied combination therapy of nasal steroid with nasal antihistamine spray (MP-AzeFlu) in people suffering from medium-to-severe allergic rhinitis. Oral rupatadine is a potent antihistamine and platelet activating factor (PAF) antagonist, which has not been studied in combination therapy in allergic rhinitis. Fluticasone propionate is a well established, first line nasal steroid.

Adults 19 years or older, seen in the Principal Investigator's office presenting with moderate-to-severe allergic rhinitis will be identified by the principal investigator and invited to participate in this prospective study. Patients will be recruited into the study in a consecutive manner. After providing consent, baseline characteristics will be collected. The investigator aims to recruit 51 patients in each study group respectively. Descriptive statistics will be used to analyze the baseline characteristic data.

ELIGIBILITY:
Inclusion Criteria:

1. Patient over the age of 18
2. Positive allergy skin prick test that diagnose AR
3. Persistent and Moderate-to-Severe AR (Persistent symptoms for more than 6 weeks and suffers from abnormal sleep, impairment of daily activities, work-school problems, or has troublesome symptoms; TNSS of at least 8/12)
4. Negative CT sinus

Exclusion Criteria:

1. Non-Allergic Rhinitis patients will be excluded from this study.
2. Participants who are pregnant or lactating
3. Hypersensitivity to FP, MP-AzeFlu, or Rupatadine
4. Superficial or moderate nasal erosion, nasal mucosal ulceration or nasal septum perforation, who had nasal surgery within the last year, had significant pulmonary disease (excluding intermittent asthma)
5. Participants who had inferior turbinate reduction surgery
6. Participants who smoke
7. Not able to read and understand the consent form
8. Patients suffering from nonallergic rhinitis (eg. vasomotor, infectious, or drug-induced rhinitis) or with a negative skin prick test will not be included

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-12-15 (Estimated); Primary Completion 2021-06-01 (Estimated); Study Completion 2021-07-01 (Estimated)

PRIMARY OUTCOMES:
Change in Reflective Total Nasal Symptom Score (TNSS) | 2 weeks
  Score range of 0 to 12, higher scores indicate worse symptoms

SECONDARY OUTCOMES:
Change in Individual reflective nasal symptoms score (iTNSS) | 2 weeks
  Score range of 0 to 12, higher scores indicate worse symptoms
Change in reflective total ocular symptoms score (rTOSS) | 2 weeks
  Score range of 0 to 12, higher scores indicate worse symptoms
Change in Rhinoconjunctivitis Quality of Life Questionnaire (RQLQ) | 6 weeks
  Score range of 0 to 168, split into 7 sections, higher the score relates to more negative impact on QoL
Adverse Events | 2 weeks
  Patient reported adverse events